CLINICAL TRIAL: NCT00790569
Title: Varenicline Versus Nicotine Replacement for Methadone-Maintained Smokers
Brief Title: Varenicline or Nicotine Patch and Nicotine Gum in Helping Smokers in a Methadone Treatment Program Stop Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael Stein, MD, Principal Investigator, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CDR0000616663; R01CA129226 (NIH); BUTLER-0807-004
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Bladder Cancer; Cervical Cancer; Esophageal Cancer; Gastric Cancer; Head and Neck Cancer; Kidney Cancer; Leukemia; Liver Cancer; Lung Cancer; Pancreatic Cancer; Tobacco Use Disorder
Keywords: bladder cancer; cervical cancer; esophageal cancer; gastric cancer; renal cell carcinoma; adult primary liver cancer; non-small cell lung cancer; small cell lung cancer; pancreatic cancer; hypopharyngeal cancer; laryngeal cancer; lip and oral cavity cancer; nasopharyngeal cancer; oropharyngeal cancer; paranasal sinus and nasal cavity cancer; adult acute myeloid leukemia; tobacco use disorder
MeSH Terms: conditions — Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Kidney Neoplasms; Leukemia; Liver Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Tobacco Use Disorder; Carcinoma, Renal Cell; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Leukemia, Myeloid, Acute | interventions — Nicotine; Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Experimental): Patients receive oral varenicline once daily on days 1-3 and twice daily thereafter for a total of 6 months or when a comfortable level of smoking abstinence is reached.
  Interventions: Drug: varenicline
- Arm II (Placebo Comparator): Patients receive oral varenicline placebo once daily on days 1-3 and twice daily thereafter for a total of 6 months or when a comfortable level of smoking abstinence is reached.
  Interventions: Other: placebo
- Arm III (Active Comparator): Patients receive a nicotine patch, with doses tapering over time for a total of 26 weeks. Patients also receive nicotine gum to quell breakthrough urges. Patients may stop treatment when a comfortable level of smoking abstinence is reached.
  Interventions: Drug: nicotine

INTERVENTIONS:
Drug: nicotine — Given transdermally and orally
  Arms: Arm III
Drug: varenicline — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Varenicline, the nicotine patch, and nicotine gum help people stop smoking. It is not yet known whether varenicline is more effective than the nicotine patch given together with nicotine gum in helping smokers quit smoking.

PURPOSE: This randomized clinical trial is studying varenicline to see how well it works compared with the nicotine patch given together with nicotine gum in helping smokers in a methadone treatment program stop smoking.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether varenicline, a nicotine receptor partial agonist, leads to a higher rate of smoking cessation than combination nicotine replacement therapy with nicotine patch prescription plus ad libitum nicotine gum delivery in methadone-maintained smokers.

Secondary

* To test the effects of the treatments on smoking urges, withdrawal symptoms, and reinforcing effects of smoking.
* To test the effects of the treatments on methadone treatment outcomes, including retention in methadone maintenance, methadone dose changes, and continued use of illicit drugs as measured by urine toxicologies.

OUTLINE: This is a multicenter study. Patients are stratified based on gender and level of nicotine dependence. Patients are randomized to 1 of 3 intervention arms.

At baseline, all patients receive a minimal behavioral intervention using a 3-minute, simple smoking cessation counseling strategy, a self-help manual, and a telephone quit-line number.

* Arm I (varenicline): Patients receive oral varenicline once daily on days 1-3 and twice daily thereafter for a total of 6 months or when a comfortable level of smoking abstinence is reached.
* Arm II (placebo): Patients receive oral varenicline placebo once daily on days 1-3 and twice daily thereafter for a total of 6 months or when a comfortable level of smoking abstinence is reached.
* Arm III (nicotine patch/gum): Patients receive a nicotine patch, with doses tapering over time for a total of 26 weeks. Patients also receive nicotine gum to quell breakthrough urges. Patients may stop treatment when a comfortable level of smoking abstinence is reached.

Patients complete a brief interview over 10-15 minutes at 2 weeks and monthly during months 1-5. They complete a longer interview over 45 minutes at months 6 and 12 and provide breath samples (for carbon monoxide monitoring) and urine samples (for cotinine testing).

NOTE: Smoking cessation may prevent certain smoking-related illnesses, including cancer.

PROJECTED ACCRUAL: A total of 602 patients (258 receiving varenicline, 258 receiving nicotine replacement therapy, and 86 receiving placebo) will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA

* Current and regular cigarette smokers (over 10 cigarettes/day for the past 3 months)
* Interested in quitting smoking

  * Willing to set a quit date 7 days after baseline assessment
* Participating in 1 of 5 methadone maintenance treatment programs across Rhode Island at any of the following institutions:

  * Codac, Inc. (with two independent sites)
  * Addiction Recovery Institute
  * Center for Treatment and Recovery
  * Discovery House
* Has received methadone for at least the past month

EXCLUSION CRITERIA

* Pregnant or nursing (Must have negative pregnancy test)
* Non-English speaking
* No personal telephone or does not live close to a relative or neighbor with a telephone
* Unwilling to make their methadone dose and methadone maintenance treatment program urine toxicologies available for review
* Unvailable for this study for the next 12 months
* Suffering from any unstable medical condition which would preclude the use of the nicotine patch (e.g., unstable angina or uncontrolled hypertension)
* Active skin condition (e.g., psoriasis)
* History of skin allergy
* History of a suicide attempt
* Working as pilots, drivers, or operators of heavy machinery

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent insulin or blood thinners
* No concurrent smokeless tobacco, nicotine replacement therapy, or other smoking cessation treatment

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2008-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stein, MD, Study Chair — Butler Hospital
Locations (1):
- Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island, United States

REFERENCES:
- [Background] Stein MD, Caviness CM, Kurth ME, Audet D, Olson J, Anderson BJ. Varenicline for smoking cessation among methadone-maintained smokers: a randomized clinical trial. Drug Alcohol Depend. 2013 Dec 1;133(2):486-93. doi: 10.1016/j.drugalcdep.2013.07.005. Epub 2013 Aug 14. PMID 23953658
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] de Dios MA, Anderson BJ, Caviness CM, Stein M. Intimate partner violence among individuals in methadone maintenance treatment. Subst Abus. 2014;35(2):190-3. doi: 10.1080/08897077.2013.835764. PMID 24821357
- [Derived] Caviness CM, Bird JL, Anderson BJ, Abrantes AM, Stein MD. Minimum recommended physical activity, and perceived barriers and benefits of exercise in methadone maintained persons. J Subst Abuse Treat. 2013 Apr;44(4):457-62. doi: 10.1016/j.jsat.2012.10.002. Epub 2012 Nov 28. PMID 23199641

RESULTS

PARTICIPANT FLOW:
Period: End of Treatment (6 Month Interview)
Arm/Group | Arm I | Arm II | Arm III
Started | 137 | 45 | 133
Completed | 115 | 35 | 107
Not Completed | 22 | 10 | 26
Not completed — Lost to Follow-up | 20 | 8 | 20
Not completed — Death | 0 | 2 | 1
Not completed — Hospitalized | 2 | 0 | 0
Not completed — Residential Treatment | 0 | 0 | 2
Not completed — Incarcerated | 0 | 0 | 3
Period: End of Study (12 Month Interview)
Arm/Group | Arm I | Arm II | Arm III
Started | 137 | 45 | 133
Completed | 71 | 26 | 83
Not Completed | 66 | 19 | 50
Not completed — Lost to Follow-up | 66 | 19 | 50

BASELINE CHARACTERISTICS:
Population: All eligible participants who completed enrollment and were randomized were included in baseline analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Arm III | Total
Number analyzed (Participants) | 137 | 45 | 133 | 315
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (9.7) | 40.6 (10.6) | 40.3 (9.3) | 39.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 17 | 68 | 159
  Male | 63 | 28 | 65 | 156
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 3 | 8
  White | 113 | 34 | 103 | 250
  More than one race | 5 | 4 | 10 | 19
  Unknown or Not Reported | 17 | 4 | 17 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 4 | 17 | 38
  Not Hispanic or Latino | 120 | 41 | 116 | 277
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 137 | 45 | 133 | 315
Years of Education [Mean (Standard Deviation); unit: years] | 11.8 (2.0) | 11.4 (1.9) | 11.9 (2.2) | 11.8 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Self- Reported 7-day Abstinence
Description: Number of participants with self-reported, 7-day abstinence at 6-months
Time Frame: 6 Months
Measure: Number; unit: participants
Arm/Group | Arm I | Arm II | Arm III
Number analyzed (Participants) | 137 | 45 | 133
participants | 11 | 3 | 16

2. Primary Outcome: Carbon Monoxide (CO)-Confirmed 7-day Abstinence
Description: Number of participants reporting 7-day abstinence at 6-months, confirmed with CO measurement.
Time Frame: 6-Months
Measure: Number; unit: participants
Arm/Group | Arm I | Arm II | Arm III
Number analyzed (Participants) | 137 | 45 | 133
participants | 5 | 1 | 11

3. Primary Outcome: Rates of Smoking Cessation Continuous From First Quit Day to 6 Months
Description: Number of participants who self-reported continuous abstinence from their initial quit day (study day 14) to 6 Months
Time Frame: 6-Months
Measure: Number; unit: participants
Arm/Group | Arm I | Arm II | Arm III
Number analyzed (Participants) | 137 | 45 | 133
participants | 2 | 0 | 2

4. Primary Outcome: Self-reported 7-day Abstinence
Description: Number of participants with self-reported 7-day abstinence at 12-months
Time Frame: 12 Months
Measure: Number; unit: participants
Arm/Group | Arm I | Arm II | Arm III
Number analyzed (Participants) | 137 | 45 | 133
participants | 4 | 3 | 11

5. Primary Outcome: CO-confirmed 7-day Abstinence
Description: Number of participants reporting 7-day abstinence at 12-months, confirmed with CO measurement.
Time Frame: 12 Months
Measure: Number; unit: participants
Arm/Group | Arm I | Arm II | Arm III
Number analyzed (Participants) | 137 | 45 | 133
participants | 4 | 1 | 8

6. Secondary Outcome: Change in Smoking Urges
Description: Smoking urges was measured on a 0 (not at all) - 100 (strongest feeling possible) scale. Higher values represent greater urge to smoke. Change in smoking urges was calculated as Follow-up score (6 month) - Baseline Score.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I | Arm II | Arm III
Number analyzed (Participants) | 89 | 26 | 86
units on a scale | -29.971 (39.120) | -25.015 (31.689) | -24.177 (37.015)

7. Secondary Outcome: Withdrawal Symptoms
Description: Withdrawal Symptoms were measured using a modified version of the Minnesota Behavior Rating Scale. The scale asked subjects to rate their smoking withdrawal symptoms over the previous 24 hours on a scale from 0 (none) to 4 (severe). Higher values indicate more severe withdrawal symptoms. Change in withdrawal symptoms was calculated as Follow-up score (6 month) - Baseline Score.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I | Arm II | Arm III
Number analyzed (Participants) | 88 | 26 | 86
units on a scale | -.222 (.618) | -.163 (.447) | -.113 (.564)

8. Secondary Outcome: Retention in Methadone Maintenance
Time Frame: 12 months
Population: Data not collected
Arm/Group | Arm I | Arm II | Arm III
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Methadone Dose Changes
Time Frame: 12 months
Population: Data not collected
Arm/Group | Arm I | Arm II | Arm III
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Use of Illicit Drugs as Measured by Urine Toxicologies
Time Frame: 12 months
Population: Data not collected
Arm/Group | Arm I | Arm II | Arm III
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Reinforcing Effects of Smoking
Description: Reinforcing effects of smoking was measured using the modified version of the Cigarette Evaluation Questionnaire. Participants were asked to indicate on a 12-item scale how smoking made them feel in the prior 30 days on a scale from 1 (Not at all) to 7 (Extremely). Higher values indicated that smoking was a more positive experience for 10 of 12 items. Two items were reverse coded. Change in reinforcing effects of smoking was calculated as Follow-up score (6 month) - Baseline Score.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I | Arm II | Arm III
Number analyzed (Participants) | 81 | 25 | 75
units on a scale | -1.005 (1.173) | -.683 (.865) | -.761 (.957)

12. Secondary Outcome: Change in Cigarettes Per Day
Description: Change in mean cigarettes per day
Time Frame: 6-Months
Measure: Mean (Standard Deviation); unit: cigarettes/day
Arm/Group | Arm I | Arm II | Arm III
Number analyzed (Participants) | 137 | 45 | 133
cigarettes/day | -8.7 (9.2) | -8.5 (9.5) | -7.8 (9.4)

ADVERSE EVENTS:
Arm/Group | Arm I | Arm II | Arm III
Serious Adverse Events (participants affected / at risk) | 4/137 | 2/45 | 2/133
Other Adverse Events (participants affected / at risk) | 0/137 | 0/45 | 0/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=137) | Arm II (N=45) | Arm III (N=133)
Neurobehavioral Adverse Effects (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Participant described hearing voices
Neurobehavioral Adverse Events (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Participant reported mood disturbance
Participant Death (General disorders) | 0 (0) | 2 (2) | 1 (1) — Participant died during study participation
Heart Attack (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Participant was hospitalized with symptoms of heat attack
Skin Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) — Participants complained of skin rashes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No